CLINICAL TRIAL: NCT05654441
Title: Low-grade Inflammatory Challenge and Social Behavior
Brief Title: Body and Social Behavior
Acronym: BSB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-1024; 2047344 (Other: National Science Foundation)
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-07

CONDITIONS: Psychology, Social; Inflammation; Defeat, Social; Interaction, Social
MeSH Terms: conditions — Inflammation; Social Defeat | interventions — Influenza Vaccines; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Influenza Vaccine (Experimental): Experimental group given influenza vaccine (Flulaval)
  Interventions: Biological: Influenza vaccine
- Sham Vaccine (Placebo Comparator): The control group given a placebo (saline injection)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Influenza vaccine — 0.5 mL single-dose injection
  Arms: Influenza Vaccine
Biological: Placebo — 0.5 mL single-dose injection with no therapeutic effect
  Other Names: Saline Injection
  Arms: Sham Vaccine

SUMMARY:
This randomized, double-blind, placebo-controlled study of the influenza vaccine will shed important light on how the immune system responds to different positive and negative social experiences. Building on the nuanced animal literature showing that, while animals exposed to an inflammatory challenge show reductions in social exploration consistent with the sickness behavior of social withdrawal, they actually show increases in social engagement behavior during interactions with a cage mate or pair-bonded animal. The present study will examine if a mild inflammatory challenge (receipt of the influenza vaccine) leads to change in actual social behavior in interactions, specifically toward a stranger and separately, toward a close friend. This study will also build on foundational animal research showing that an inflammatory challenge leads to social defeat behaviors in animals.

DETAILED DESCRIPTION:
Psychologists have long appreciated that the mind can impact the body, and that bodily changes can influence the mind. Social psychologists in particular have conducted pioneering work on connections between the mind and body, showing both that social experiences elicit changes in numerous physiological systems and that physiological changes influence social cognition and behavior. Until recently, however, little attention has been paid to the connections between social experiences and the immune system. This is a critical gap knowledge, as seminal animal work shows that there are profound relationships between social experiences and immune system functioning that have yet to be fully explored in humans. Further, there are strong theoretical reasons to suspect that the immune system matters for social psychological processes even beyond times of sickness, though many of these connections are yet to be uncovered empirically in humans. Thus, to develop a comprehensive understanding of the mind-body connections that drive social behavior, researchers must integrate the immune system.

To address this critical gap in knowledge, the present study will examine the body-to-mind connection between the immune system and positive (i.e., interacting with a close other) and negative (i.e., social defeat) social experiences.

Why does the immune system matter for social behavior? There are good theoretical reasons why the immune system would be tightly interconnected to even normative, everyday social experiences beyond times of sickness. First, despite the common belief that the immune system only comes "online" in response to pathogens or physical injury, the immune system is in fact always active and fluctuates considerably even in the absence of an acute infection. Indeed, the immune system is responsive to both real and imagined situations that may signal increased probability of injury or infection. This includes everyday social experiences and situations of greater interest to social psychologists, from falling in love to being socially ostracized. Second, the brain is constantly monitoring the physiological state of the body and integrating this interoceptive information with signals from the broader environment to anticipate current and future metabolic demands and guide adaptive behavior. Thus, even relatively minor fluctuations in immune system activation beyond times of sickness can feed back to the brain to guide social cognition and behavior. In sum, there are strong theoretical reasons why everyday, normative social experiences may affect and be affected by immune system activation.

To date, social withdrawal is considered a hallmark "sickness behavior", based on both animal and human work showing that experimentally-induced increases in inflammation lead to less social exploration and greater feelings of social disconnection. However, other animal work suggests that the effects of inflammation on social behavior may be more nuanced than uniform social withdrawal, as some research shows that animals spend more time huddling with familiar cagemates, and form pair bonds more quickly when exposed to an inflammatory challenge. Further, recent work in the field of psychoneuroimmunology with humans replicates this, showing that an inflammatory challenge causes heightened (not diminished) neural responses to reminders of social connection. Yet to date, no known human work has examined if an inflammatory challenge causes changes in actual social behavior in humans, a critical next step in this line of research. Techniques from experimental social psychology are ideally-suited to address this next step, as social psychology has been at the cutting-edge of developing tools for eliciting and quantifying social behavior, particularly in the context of dyadic interactions that are likely to be important during an inflammatory challenge. This study will bring this important perspective to bear to further understanding of how immune system activation may cause changes in social behavior.

There is a storied history in psychoneuroimmunology (PNI) of using vaccines (e.g., influenza, typhoid) as a way to study immune system functioning. In vaccine trials, researchers typically examine how individual-differences in psychological processes (e.g., depressive symptoms, social connection) influence the effectiveness of the vaccine by examining the number of antibody titers produced following vaccination as a function of the individual-difference of interest. More recently, researchers have begun to use the influenza vaccine as a way to manipulate levels of inflammation, as the vaccine produces a small, but significant, increase in inflammatory markers (e.g., interleukin-6) in the 24-hours following vaccination administration. Prior work has examined the impact of vaccine-induced increases in inflammation on psychological processes such as mood and reward processing and shown that within-subject changes in inflammation in response to the influenza vaccine predict increases in daily negative affect and increases in reward responsivity. The present project will build on this prior work by adding a placebo-controlled (saline) condition, thus allowing researchers to determine if vaccine-induced changes in inflammation cause changes in social behavior. Using the influenza vaccine as an inflammatory challenge has numerous advantages over prior approaches: 1) It provides a public health service to the local community (i.e., given that vaccinations can prevent viral outbreaks) rather than making participants temporarily ill, as in the rhinovirus studies and endotoxin studies discussed previously; 2) The change in inflammation elicited by the vaccine is relatively small, thus mirroring more normative, day-to-day fluctuations in inflammation beyond times of sickness; and 3) Experimental procedures are less resource and cost-intensive, as almost every local pharmacy provides influenza vaccinations, and the cost is often covered by insurance and is relatively low (or free) for the uninsured. Given these advantages, the present study will use the influenza vaccine to examine if an experimental manipulation of inflammation causes changes in social behavior of interest to both social psychologists and psychoneuroimmunologists. In doing so, the study will advance a method that can be widely adopted by researchers to study how immune system activation feeds back to the brain to influence social experience.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Have a same-gender friend willing to participate in the second study session

Exclusion Criteria:

* Are not a student
* Have already received the annual influenza vaccine or had the flu this season
* Report current illness/sickness symptoms, including upper respiratory symptoms
* Report any major medical conditions (e.g., diabetes, asthma)
* Use mood or immune altering medications (e.g., anti-depressants)
* Current regular nicotine/tobacco use (i.e., daily use of cigarettes or e-cigarettes)
* Have an allergy to eggs
* Have had COVID-19 in past two weeks
* Current or history of depression or anxiety
* Have had Guillain-Barre Syndrome
* Are allergic to vaccine or ingredients present in vaccine
* Have had an adverse reaction to a blood draw, including to needles or sight or blood
* Weigh less than 110 pounds
* Are unwilling to be video/audio recorded during the social interaction tasks
* Are unwilling to be unmasked during the social interaction tasks

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keely Muscatell, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Clinical and Translation Research Center, Chapel Hill, North Carolina
  - Howell Hall, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning immediately following publication and ending 5 years after article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Barrett LF. The theory of constructed emotion: an active inference account of interoception and categorization. Soc Cogn Affect Neurosci. 2017 Jan 1;12(1):1-23. doi: 10.1093/scan/nsw154. PMID 27798257
- [Background] SCHACHTER S, SINGER JE. Cognitive, social, and physiological determinants of emotional state. Psychol Rev. 1962 Sep;69:379-99. doi: 10.1037/h0046234. No abstract available. PMID 14497895
- [Background] Dickerson SS, Kemeny ME. Acute stressors and cortisol responses: a theoretical integration and synthesis of laboratory research. Psychol Bull. 2004 May;130(3):355-91. doi: 10.1037/0033-2909.130.3.355. PMID 15122924
- [Background] Richeson JA, Shelton JN. Negotiating Interracial Interactions: Costs, Consequences, and Possibilities. Current Directions in Psychological Science. 2007;16(6):316-320. doi:10.1111/j.1467-8721.2007.00528.x
- [Background] Siegel EH, Sands MK, Van den Noortgate W, Condon P, Chang Y, Dy J, Quigley KS, Barrett LF. Emotion fingerprints or emotion populations? A meta-analytic investigation of autonomic features of emotion categories. Psychol Bull. 2018 Apr;144(4):343-393. doi: 10.1037/bul0000128. Epub 2018 Feb 1. PMID 29389177
- [Background] Bartz JA, Zaki J, Bolger N, Ochsner KN. Social effects of oxytocin in humans: context and person matter. Trends Cogn Sci. 2011 Jul;15(7):301-9. doi: 10.1016/j.tics.2011.05.002. Epub 2011 Jun 21. PMID 21696997
- [Background] Storbeck J, Clore GL. Affective Arousal as Information: How Affective Arousal Influences Judgments, Learning, and Memory. Soc Personal Psychol Compass. 2008 Sep 1;2(5):1824-1843. doi: 10.1111/j.1751-9004.2008.00138.x. PMID 25067943
- [Background] Eisenberger NI, Moieni M, Inagaki TK, Muscatell KA, Irwin MR. In Sickness and in Health: The Co-Regulation of Inflammation and Social Behavior. Neuropsychopharmacology. 2017 Jan;42(1):242-253. doi: 10.1038/npp.2016.141. Epub 2016 Aug 2. PMID 27480575
- [Background] Gassen J, Hill SE. Why inflammation and the activities of the immune system matter for social and personality psychology (and not only for those who study health). Soc Personal Psychol Compass. May 2019:e12471. doi:10.1111/spc3.12471
- [Background] Kemeny ME. Psychobiological responses to social threat: evolution of a psychological model in psychoneuroimmunology. Brain Behav Immun. 2009 Jan;23(1):1-9. doi: 10.1016/j.bbi.2008.08.008. Epub 2008 Sep 10. PMID 18809488
- [Background] Hennessy MB, Deak T, Schiml PA. Sociality and sickness: have cytokines evolved to serve social functions beyond times of pathogen exposure? Brain Behav Immun. 2014 Mar;37:15-20. doi: 10.1016/j.bbi.2013.10.021. Epub 2013 Oct 31. PMID 24184399
- [Background] Dhabhar FS, Malarkey WB, Neri E, McEwen BS. Stress-induced redistribution of immune cells--from barracks to boulevards to battlefields: a tale of three hormones--Curt Richter Award winner. Psychoneuroendocrinology. 2012 Sep;37(9):1345-68. doi: 10.1016/j.psyneuen.2012.05.008. Epub 2012 Jun 22. PMID 22727761
- [Background] Leschak CJ, Eisenberger NI. Two Distinct Immune Pathways Linking Social Relationships With Health: Inflammatory and Antiviral Processes. Psychosom Med. 2019 Oct;81(8):711-719. doi: 10.1097/PSY.0000000000000685. PMID 31600173
- [Background] Slavich GM, Irwin MR. From stress to inflammation and major depressive disorder: a social signal transduction theory of depression. Psychol Bull. 2014 May;140(3):774-815. doi: 10.1037/a0035302. Epub 2014 Jan 13. PMID 24417575
- [Background] Slavich GM, Cole SW. The Emerging Field of Human Social Genomics. Clin Psychol Sci. 2013 Jul;1(3):331-348. doi: 10.1177/2167702613478594. PMID 23853742
- [Background] Murray DR, Haselton MG, Fales M, Cole SW. Falling in love is associated with immune system gene regulation. Psychoneuroendocrinology. 2019 Feb;100:120-126. doi: 10.1016/j.psyneuen.2018.09.043. Epub 2018 Oct 2. PMID 30299259
- [Background] Muscatell KA, Dedovic K, Slavich GM, Jarcho MR, Breen EC, Bower JE, Irwin MR, Eisenberger NI. Greater amygdala activity and dorsomedial prefrontal-amygdala coupling are associated with enhanced inflammatory responses to stress. Brain Behav Immun. 2015 Jan;43:46-53. doi: 10.1016/j.bbi.2014.06.201. Epub 2014 Jul 9. PMID 25016200
- [Background] Slavich GM, Way BM, Eisenberger NI, Taylor SE. Neural sensitivity to social rejection is associated with inflammatory responses to social stress. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14817-22. doi: 10.1073/pnas.1009164107. Epub 2010 Aug 2. PMID 20679216
- [Background] Sterling P. Allostasis: a model of predictive regulation. Physiol Behav. 2012 Apr 12;106(1):5-15. doi: 10.1016/j.physbeh.2011.06.004. Epub 2011 Jun 12. PMID 21684297
- [Background] Dantzer R, O'Connor JC, Freund GG, Johnson RW, Kelley KW. From inflammation to sickness and depression: when the immune system subjugates the brain. Nat Rev Neurosci. 2008 Jan;9(1):46-56. doi: 10.1038/nrn2297. PMID 18073775
- [Background] Hart BL. Biological basis of the behavior of sick animals. Neurosci Biobehav Rev. 1988 Summer;12(2):123-37. doi: 10.1016/s0149-7634(88)80004-6. PMID 3050629
- [Background] Avitsur R, Cohen E, Yirmiya R. Effects of interleukin-1 on sexual attractivity in a model of sickness behavior. Physiol Behav. 1997 Dec 31;63(1):25-30. doi: 10.1016/s0031-9384(97)00381-8. PMID 9402610
- [Background] Bluthe RM, Dantzer R, Kelley KW. Effects of interleukin-1 receptor antagonist on the behavioral effects of lipopolysaccharide in rat. Brain Res. 1992 Feb 28;573(2):318-20. doi: 10.1016/0006-8993(92)90779-9. PMID 1387028
- [Background] Eisenberger NI, Inagaki TK, Mashal NM, Irwin MR. Inflammation and social experience: an inflammatory challenge induces feelings of social disconnection in addition to depressed mood. Brain Behav Immun. 2010 May;24(4):558-63. doi: 10.1016/j.bbi.2009.12.009. Epub 2010 Jan 4. PMID 20043983
- [Background] Moieni M, Irwin MR, Jevtic I, Olmstead R, Breen EC, Eisenberger NI. Sex differences in depressive and socioemotional responses to an inflammatory challenge: implications for sex differences in depression. Neuropsychopharmacology. 2015 Jun;40(7):1709-16. doi: 10.1038/npp.2015.17. Epub 2015 Jan 19. PMID 25598426
- [Background] Willette AA, Lubach GR, Coe CL. Environmental context differentially affects behavioral, leukocyte, cortisol, and interleukin-6 responses to low doses of endotoxin in the rhesus monkey. Brain Behav Immun. 2007 Aug;21(6):807-15. doi: 10.1016/j.bbi.2007.01.007. Epub 2007 Mar 1. PMID 17336039
- [Background] Yee JR, Prendergast BJ. Sex-specific social regulation of inflammatory responses and sickness behaviors. Brain Behav Immun. 2010 Aug;24(6):942-51. doi: 10.1016/j.bbi.2010.03.006. Epub 2010 Mar 17. PMID 20303405
- [Background] Bilbo SD, Klein SL, DeVries AC, Nelson RJ. Lipopolysaccharide facilitates partner preference behaviors in female prairie voles. Physiol Behav. 1999 Dec 1-15;68(1-2):151-6. doi: 10.1016/s0031-9384(99)00154-7. PMID 10627074
- [Background] Inagaki TK, Muscatell KA, Irwin MR, Moieni M, Dutcher JM, Jevtic I, Breen EC, Eisenberger NI. The role of the ventral striatum in inflammatory-induced approach toward support figures. Brain Behav Immun. 2015 Feb;44:247-52. doi: 10.1016/j.bbi.2014.10.006. Epub 2014 Oct 16. PMID 25459101
- [Background] Muscatell KA, Moieni M, Inagaki TK, Dutcher JM, Jevtic I, Breen EC, Irwin MR, Eisenberger NI. Exposure to an inflammatory challenge enhances neural sensitivity to negative and positive social feedback. Brain Behav Immun. 2016 Oct;57:21-29. doi: 10.1016/j.bbi.2016.03.022. Epub 2016 Mar 28. PMID 27032568
- [Background] Aron A, Melinat E, Aron EN, Vallone RD, Bator RJ. The Experimental Generation of Interpersonal Closeness: A Procedure and Some Preliminary Findings. Pers Soc Psychol Bull. 1997;23(4):363-377. doi:10.1177/0146167297234003
- [Background] Berger J, Heinrichs M, von Dawans B, Way BM, Chen FS. Cortisol modulates men's affiliative responses to acute social stress. Psychoneuroendocrinology. 2016 Jan;63:1-9. doi: 10.1016/j.psyneuen.2015.09.004. Epub 2015 Sep 5. PMID 26398000
- [Background] Glaser R, Robles TF, Sheridan J, Malarkey WB, Kiecolt-Glaser JK. Mild depressive symptoms are associated with amplified and prolonged inflammatory responses after influenza virus vaccination in older adults. Arch Gen Psychiatry. 2003 Oct;60(10):1009-14. doi: 10.1001/archpsyc.60.10.1009. PMID 14557146
- [Background] Pressman SD, Cohen S, Miller GE, Barkin A, Rabin BS, Treanor JJ. Loneliness, social network size, and immune response to influenza vaccination in college freshmen. Health Psychol. 2005 May;24(3):297-306. doi: 10.1037/0278-6133.24.3.297. PMID 15898866
- [Background] Christian LM, Iams JD, Porter K, Glaser R. Inflammatory responses to trivalent influenza virus vaccine among pregnant women. Vaccine. 2011 Nov 8;29(48):8982-7. doi: 10.1016/j.vaccine.2011.09.039. Epub 2011 Sep 22. PMID 21945263
- [Background] Tsai MY, Hanson NQ, Straka RJ, Hoke TR, Ordovas JM, Peacock JM, Arends VL, Arnett DK. Effect of influenza vaccine on markers of inflammation and lipid profile. J Lab Clin Med. 2005 Jun;145(6):323-7. doi: 10.1016/j.lab.2005.03.009. PMID 15976761
- [Background] Boyle CC, Kuhlman KR, Dooley LN, Haydon MD, Robles TF, Ang YS, Pizzagalli DA, Bower JE. Inflammation and dimensions of reward processing following exposure to the influenza vaccine. Psychoneuroendocrinology. 2019 Apr;102:16-23. doi: 10.1016/j.psyneuen.2018.11.024. Epub 2018 Nov 20. PMID 30496908
- [Background] Kuhlman KR, Robles TF, Dooley LN, Boyle CC, Haydon MD, Bower JE. Within-subject associations between inflammation and features of depression: Using the flu vaccine as a mild inflammatory stimulus. Brain Behav Immun. 2018 Mar;69:540-547. doi: 10.1016/j.bbi.2018.02.001. Epub 2018 Feb 16. PMID 29458196
- [Background] Kuhlman KR, Robles TF, Haydon MD, Dooley L, Boyle CC, Bower JE. Early life stress sensitizes individuals to the psychological correlates of mild fluctuations in inflammation. Dev Psychobiol. 2020 Apr;62(3):400-408. doi: 10.1002/dev.21908. Epub 2019 Sep 6. PMID 31489628

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Influenza Vaccine | Sham Vaccine
Started | 52 | 52
Completed | 52 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine | Sham Vaccine | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.46 (1.69) | 20.62 (2.61) | 20.54 (2.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 77
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 47 | 46 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 10 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 31 | 27 | 58
  More than one race | 3 | 7 | 10
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 50 | 102

OUTCOME MEASURES:

1. Primary Outcome: IL-6 Levels 24 Hours After Vaccine
Description: The investigators will examine levels of IL-6 measured in plasma 24-hours following the vaccine.
Time Frame: within approximately 24 hours of treatment
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Measure: Mean (Standard Deviation); unit: log pg/mL
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
log pg/mL | 0.40 (0.25) | 0.23 (0.23)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p < 0.001, ANOVA

2. Primary Outcome: IL-10 Levels 24 Hours After Vaccine
Description: The investigators will examine levels of IL-10 measured in plasma 24-hours following the vaccine.
Time Frame: within approximately 24 hours of treatment
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Measure: Mean (Standard Deviation); unit: log pg/mL
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
log pg/mL | 0.50 (0.14) | 0.36 (0.14)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p < 0.001, ANOVA

3. Primary Outcome: TNF-alpha Levels 24 Hours After Vaccine
Description: The investigators will examine levels of TNF-alpha measured in plasma 24-hours following the vaccine.
Time Frame: within approximately 24 hours of treatment
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Measure: Mean (Standard Deviation); unit: log pg/mL
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
log pg/mL | 0.93 (0.10) | 0.88 (0.10)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p = 0.007, ANOVA

4. Primary Outcome: IFN-gamma Levels 24 Hours After Vaccine
Description: The investigators will examine levels of IFN-gamma measured in plasma 24-hours following the vaccine.
Time Frame: within approximately 24 hours of treatment
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Measure: Mean (Standard Deviation); unit: log pg/mL
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
log pg/mL | 0.44 (0.38) | -0.14 (0.21)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p < 0.001, ANOVA

5. Secondary Outcome: Sickness Symptom Scores
Description: The investigators will examine if there are differences in self-reported sickness symptoms, as measured by the Sickness Questionnaire, as a function of vaccine condition. The 10-item Sickness Questionnaire includes Likert-type questions using a 4- point scale, the total range is 0-30 with higher scores indicating greater sickness symptoms.
Time Frame: within approximately 24 hours of treatment
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
score on a scale | 7.00 (4.39) | 7.12 (4.12)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p = 0.886, t-test, 2 sided

6. Secondary Outcome: High Arousal Negative Affect Scores
Description: he investigators will examine if there are differences in self-reported high arousal negative affect, as measured by a subscale of the Positive Affect-Negative Affect Schedule-X, as a function of vaccine condition. Participants indicated the extent to which they felt each of 11 high arousal negative emotions (i.e., "angry", "irritable", "nervous", "scared", "upset", "afraid", "ashamed", "distressed", "frustrated", "hostile", "jittery") on a 0 (not at all) -100 (extremely) sliding scale. Responses were then averaged with higher scores indicating greater high arousal negative affect.
Time Frame: within approximately 24 hours of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
score on a scale | 8.67 (11.94) | 7.64 (11.95)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p = .666, t-test, 2 sided

7. Secondary Outcome: Low Arousal Negative Affect Scores
Description: The investigators will examine if there are differences in self-reported low arousal negative affect, as measured by a subscale of the Positive Affect-Negative Affect Schedule-X, as a function of vaccine condition. Participants indicated the extent to which they felt each of four low arousal negative emotions (i.e., "bored", "guilty", "sad", "worn out") on a 0 (not at all) -100 (extremely) sliding scale. Responses were then averaged with higher scores indicating greater low arousal negative affect.
Time Frame: within approximately 24 hours of treatment
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
score on a scale | 20.35 (16.02) | 18.19 (16.02)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p = .522, t-test, 2 sided

8. Secondary Outcome: High Arousal Positive Affect Scores
Description: The investigators will examine if there are differences in self-reported high arousal positive affect, as measured by a subscale of the Positive Affect-Negative Affect Schedule-X, as a function of vaccine condition. Participants indicated the extent to which they felt each of 10 high arousal positive emotions (i.e., "amused," "determined," "enthusiastic," "excited," "happy," "inspired", "proud," "strong," "active," "alert") on a 0 (not at all) -100 (extremely) sliding scale. Responses were then averaged with higher scores indicating greater high arousal positive affect.
Time Frame: within approximately 24 hours of treatment
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
score on a scale | 37.30 (20.54) | 33.99 (22.12)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p = .438, t-test, 2 sided

9. Secondary Outcome: Low Arousal Positive Affect Scores
Description: The investigators will examine if there are differences in self-reported low arousal positive affect, as measured by a subscale of the Positive Affect-Negative Affect Schedule-X, as a function of vaccine condition. Participants indicated the extent to which they felt each of 5 low arousal positive emotions (i.e., "attentive," "calm", "interested", "grateful", "relieved") on a 0 (not at all) -100 (extremely) sliding scale. Responses were then averaged with higher scores indicating greater low arousal positive affect.
Time Frame: within approximately 24 hours of treatment
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
score on a scale | 48.71 (18.83) | 43.50 (20.06)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p = .181, t-test, 2 sided

10. Secondary Outcome: Sleep Quality Scores
Description: The investigators will examine if there are differences in self-reported sleep quality, as measured by five items adapted from the Brief Pittsburgh Sleep Quality Index, as a function of vaccine condition. The 5-item scale assess sleep duration, sleep quality, daytime dysfunction, sleep latency, and nighttime disturbances- each producing a score ranging from 0 to 3. These scores are then summed; the total range is 0-15 with higher scores indicating poorer sleep.
Time Frame: within approximately 24 hours of treatment
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
score on a scale | 5.13 (2.23) | 5.13 (2.23)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p = .833, t-test, 2 sided

11. Secondary Outcome: Social Disconnection Scores
Description: The investigators will examine if there are differences in self-reported social disconnection, as measured by a subset of items utilized in prior research (Moieni et al., 2015), as a function of vaccine condition. The 10-item scale includes Likert-type questions using a 5- point scale ranging from 1 (Not at all) to 5 (Very much so) which are then averaged; the total range is 0-5 with higher scores indicating greater feelings of social disconnection.
Time Frame: within approximately 24 hours of treatment
Population: Two Sham vaccine participants were excluded from analyses due to use of hydroxyzine before session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Influenza Vaccine | Sham Vaccine
Number analyzed (Participants) | 52 | 50
score on a scale | 2.34 (.44) | 2.42 (.65)
Statistical Analysis 1: Comparison: Influenza Vaccine vs Sham Vaccine; Test type: Other; p = .455, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through ~30 hours later, after completion of study procedures
Arm/Group | Influenza Vaccine | Sham Vaccine
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT05654441/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT05654441/ICF_000.pdf